CLINICAL TRIAL: NCT00359086
Title: A Phase II Study of MGCD0103 (MG-0103) Given Three Times Weekly in Patients With Relapsed and Refractory Lymphoma
Brief Title: Study of MGCD0103 Given Three Times Weekly in Patients With Relapsed and Refractory Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-008
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Lymphoma
Keywords: Relapsed and Refractory Lymphoma; Phase II
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MGCD0103

INTERVENTIONS:
Drug: MGCD0103 — MGCD0103 given orally three times per week

SUMMARY:
In this study, MGCD0103, a new anticancer drug under investigation, is given three times weekly to patients with relapsed and refractory lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of relapsed or refractory lymphoma.

  1. DLBCL stage II-IV
  2. Follicular lymphoma
* At least one site of measurable disease (≥ 2.0 cm with conventional techniques; physical exam [PE], CT, X-ray, MRI).
* Prior treatment:

  1. DLBCL cohort: Disease progression following initial therapy and transplant (unless the patient is ineligible or refused transplant). There is no limit to number of prior therapies.
  2. Follicular lymphoma cohort: Follicular lymphoma that is relapsed following or refractory to standard therapy and/or existing therapies or are not eligible for or are unlikely to achieve clinical benefit from those therapies. Patients must have failed 3 or more prior therapies.
* Must have at least one of the following considered related to disease:

  1. Local symptoms due to progressive or bulky nodal disease.
  2. Compromise of normal organ function due to progressive or bulky disease.
  3. Presence of systemic B symptoms.
  4. Presence of symptomatic extranodal disease.
  5. Cytopenias due to extensive bone marrow infiltration, autoimmune hemolytic anemia or thrombocytopenia, or hypersplenism.
* ECOG performance status of 0 or 1.
* Aged 18 years or older.
* Laboratory requirements.

Exclusion Criteria:

* Patients with another active cancer (excluding basal cell carcinoma or cervical intraepithelial neoplasia [CIN/cervical in situ] or melanoma in situ). Prior history of cancer is allowed, as long as there is no active disease.
* Pregnant or lactating women.
* Patients with uncontrolled intercurrent illness, active or uncontrolled infections, or a fever >38.5 Celsius (not due to tumor fever) on the day of scheduled dosing.
* Patients with a history of pericardial disease.
* Patients with small, moderate or large pericardial effusions or patients with a diagnosis of pericarditis.
* Patients with significant cardiac abnormalities.
* Patients with serious illnesses, medical conditions, or other medical history which would be likely to interfere with patient's participation in the study or with the interpretation of the results.
* Patients who have been treated with any investigational drug within 28 days prior to study initiation.
* Known hypersensitivity to HDAC inhibitors and to any components of MGCD0103.
* Known human immunodeficiency virus (HIV) or active Hepatitis B or C.
* Central nervous system lymphoma and lymphoma involving leptomeningeal area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 1 year (anticipated)

SECONDARY OUTCOMES:
Progression-free survival | 1 year (anticipated)
Duration of objective response | 1 year (anticipated)
Safety profile | 1 year (anticipated)
Pharmacokinetics | 1 year (anticipated)
Pharmacodynamics | 1 year (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (5):
- United States (2):
  - Duke University Adult Bone Marrow Transplant Clinic, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Canada (3):
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Charles LeMoyne Hospital, Greenfield Park, Quebec
  - Sir Mortimer Davis-Jewish General Hospital, Montreal, Quebec